CLINICAL TRIAL: NCT02445118
Title: Local Skin and Volume Changes With the Use of Allograft Adipose Matrix (AAM) in the Subcutaneous Human Dorsal Wrist, a Pilot Study
Brief Title: Allograft Adipose Matrix (AAM) in Subcutaneous Dorsal Wrist
Status: Completed | Type: Observational
Sponsor: Musculoskeletal Transplant Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: MTF 184N
Record Dates: First submitted 2015-03-25; First posted 2015-05-15 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2015-05

CONDITIONS: Aesthetic Rejuvenation
Keywords: adipose, allograft
MeSH Terms: interventions — Injections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adipose Allograft Matrix Injection: AAM injected to create a 2 to 3mm raised wheal on the proximal dorsal wrist of the non-dominant hand
  Interventions: Other: Adipose Allograft Matrix (AAM) injection

INTERVENTIONS:
Other: Adipose Allograft Matrix (AAM) injection — Adipose Allograft Matrix (AAM) injection, Non-dominant wrist

SUMMARY:
This is a 16 week pilot study to assess short term outcomes of an injectable allograft adipose matrix (AAM) in the subcutaneous space in the dorsum of the wrist. A total of 30 patients will be enrolled at 2 sites and will be followed for sixteen weeks. Volume retention and local skin changes will be observed and documented prior to and following injection at week 0 and at follow up visits at 2, 10 and 16 weeks. Evaluations will be done via photographic analysis at week 0,2,10 and 16 weeks and half of the patients will undergo magnetic resonance imaging at week zero and at week 16. The dominant wrist will serve as a control and will receive no injection. Analysis includes volume retention, tissue analysis, local skin changes and adverse events, if any.

DETAILED DESCRIPTION:
This pilot study focuses on three primary objectives: to evaluate volume retention at the site of injected allograft adipose matrix (AAM), to obtain tissue analysis via magnetic resonance imaging at the site of injection and to evaluate local skin changes as a result of the injection of AAM with follow up over a 16 week period. The AAM is derived from cadaveric human adipose recovered, processed, dehydrated and distributed by the study sponsor from thoroughly screened donors. It is distributed with instructions for rehydration prior to single use. The injection site (non-dominant wrist) will be infiltrated with Lidocaine 0.5%, Epinepherine 1:200,000 prior to AAM injection. Volume of AAM necessary to create a centered 2-3mm raised wheal at the first proximal dorsal wrist crease will be administered. Photographs taken prior and following the injection and at each of the subsequent visits are taken with a color standard within the frame for later color change analysis of the injection surrounding area. Both the control and treated hand/wrist will be photographed separately in numerous positions (extension, flexion and several degrees of either) at heart level, at week 0,2,10 and 16 weeks. A clinical assessment scale for evaluation of skin changes in appearance will also be done at these same times. Patients will be advised to avoid prolonged pressure to the dorsal wrists, wear no jewelry or wrist bands, etc., for the duration of their participation in the study. Those patients designated for MR imaging shall have their MRIs done within 3 to 5 days of their week zero and week16 visits. The images shall be read and documented by a single independent radiologist.

ELIGIBILITY:
Inclusion Criteria:

* Female,
* Between 35 and 75 years of age,
* Well controlled blood pressure,
* Able to sign an informed consent

Exclusion Criteria:

* Patients with active infection,
* Patients with a body weight change of greater than 5% throughout the 16 weeks of their participation,
* Patients with a BMI of greater than 30,
* Patients with a collagen vascular disease,
* Patients with end-stage organ failure (advanced COPD, CRF, CHF),
* Patients with lymphedema or mastectomy or axillary lymph node dissection, Patients who smoke,
* Patients that have undergone deep chemical peels, lasers, Ultherapy, Thermage, other light or energy based procedures to the dorsum of the hands one year prior,
* Patients who have taken any medication or oral supplements for the previous 4 weeks that could prolong bleeding time (e.g; Aspirin, Plavix, nutritional supplements starting with G, omega-3 , fish oil, etc)

Ages: 35 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Non-smoking females between 45 and 65 years of age with a BMI <30, with well controlled blood pressure, no active infections, collagen disorders,vascular diseases, history of lymphedema, mastectomy, lymph node dissection, end stage organ failure such as COPD, CRF, or CHF, and who have not undergone deep chemical peels, laser, Ultherapy, Thermage or other light or energy based procedures to the dorsum of the hands within the past year.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2015-05; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
2-3mm raised wheal volume retention in dorsal wrist injected with AAM at 16 weeks | 16 weeks
  Using a volume assessment scale photographs of treated vs. non-treated dorsal wrist will be evaluated by three plastic surgeons, with mean outcomes for each patient documented as final evidence

SECONDARY OUTCOMES:
Sub-Dermal Tissue Analysis | 16 weeks
  Magnetic resonance imaging taken at pre-injection (Week 0) and at 16 weeks of treated and non treated dorsal wrists will be evaluated by an independent radiologist for sub dermal adipose persistence
Local skin changes | 16 weeks
  via clinical observation and photographic evidence taken at pre-injection and at pre and post week 0, 2,10 and 16 weeks of treated and non treated dorsal wrists. local skin changes such as pore size, redness, swelling will be documented by study surgeon
Volume retention during the study interim period, documented at weeks 2 and 10 | 8 weeks
  Using a volume assessment scale, photographs of treated vs. non-treated dorsal wrist will be evaluated by three plastic surgeons, using data collected at interim time points during the study; specifically, week 2 and week 10

CONTACTS AND LOCATIONS:
Overall Officials: Sydney R. Coleman, MD, Principal Investigator — Study Principal Investigator; Roger K Khouri, MD, Principal Investigator — Study Principal Investigator
Locations (2):
- United States (2):
  - Miami Hand Center, Key Biscayne, Florida
  - Tribeca Plastic Surgery, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kokai LE, Schilling BK, Chnari E, Huang YC, Imming EA, Karunamurthy A, Khouri RK, D'Amico RA, Coleman SR, Marra KG, Rubin JP. Injectable Allograft Adipose Matrix Supports Adipogenic Tissue Remodeling in the Nude Mouse and Human. Plast Reconstr Surg. 2019 Feb;143(2):299e-309e. doi: 10.1097/PRS.0000000000005269. PMID 30688888